CLINICAL TRIAL: NCT03873207
Title: A Prospective Randomized Trial Comparing PopSole™ Offloading Device to Standard of Care Methods for the Reduction of Pain and Expedited Recovery in Patients Post Fat Graft Procedure
Brief Title: Offloading Device for Post Surgical Foot Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study (NCT03873207) was closed with the University of Pittsburgh's HRPO office (STUDY19080348) in January 2021, prior to enrolling any subjects.
Sponsor: Jeffrey A. Gusenoff, MD (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Jeffrey A. Gusenoff, MD, Professor of Plastic Surgery, University of Pittsburgh School of Medicine, Co-Director, Life After Weight Loss Program, Director, Foot Fat Grafting Institute, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19080348
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Plantar Fascitis; Fat Pad Syndrome

STUDY DESIGN:
Intervention Model Description: prospective, randomized two cohort (device or SOC) pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): Pedal fat grafting followed by PopSole™ offloading device
  Interventions: Device: PopSole™ offloading device
- Standard of care (Other): Pedal fat grafting followed by standard post-operative care with padding of the insoles
  Interventions: Device: padded insole

INTERVENTIONS:
Device: PopSole™ offloading device — Offload Device Distribution to remain in use at all times during ambulation and activity instruction to stay off of feet as much as possible for 3 days, then limit ambulation to 10 minutes per hour for 4 weeks and no sports, kicking, running or exercise for 4 weeks. Devices will be provided for both feet to maintain symmetry and gait stability between the two feet.
  Arms: Intervention
Device: padded insole — the control arm will be provided with standard padded insole to wear inside footwear
  Arms: Standard of care

SUMMARY:
Study goals are to determine if a novel post-surgical foot offloading device can reduce post-operative pain and expedite the return to daily activity following fat grafting. Investigators will perform a prospective, randomized study utilizing PopSole™, a novel fully customizable post-operative shoe insert, to aid in the recovery of patients post-surgical fat graft injections for pain and limited activity due to foot disorders (ie. fat pad atrophy of the forefoot, heel, or for chronic plantar fasciitis).

Standard of care fat grafting is often used in plastic surgery for cosmetic or reconstructive reasons. Foot fat grafting, though not considered part of this research trial, is routinely offered in the UPMC Aesthetic Plastic Surgery center as a cosmetic surgery option; however, treatment modality options following the completion of a foot fat grafting procedure to protect the fat grafts and reduce weight bearing on the fresh fat grafts are limited. Current standard of care options including crutches, scooters, bulky post-operative shoes (ie. Darco shoes [Darco Intl. Huntington WV.]), and the addition of padding to insoles or orthotics that attempt to offload the treated area. Most of these devices are flat and provide poor anatomical support, leading to compensatory gait issues which can lead to further problems and pain in the knees, hips, and back. The most common complication with post-operative foot gear is non-compliance: patients do not wear it.

The investigators have devised a novel foot offloading device (PopSole™) which will allow for customization of the area where the fat has been injected into the foot, as well as allow for customizable arch support and elevation of the metatarsals. By randomizing patients to recovery with standard methods versus this new device, the investigators are hopeful for earlier patient ambulation and return to work with decreased pain.

DETAILED DESCRIPTION:
Subjects will complete the following screening research procedures:

1. Baseline reported outcome measures (PROMs) questionnaires and surveys that will take approximately 25 minutes to complete:

   * Foot and Ankle Ability Measure (FAAM) questionnaire to assess subject ADL and function ability
   * Mayo Clinical Scoring System questionnaire (MAYO) to assess subject pain, activity and function
   * American Orthopaedic Foot and Ankle Society questionnaire (AOFAS) to assess subject pain and function
   * Manchester Foot and Ankle Disability Index to assess subject foot pain/discomfort
   * Pittsburgh Foot Survey to assess subject pain, activity, life satisfaction/quality of life
   * Offload Device Survey to assess the ease and comfort of the offload device
2. Foot ultrasounds will be performed to assess and measure baseline thickness of the plantar fascia, forefoot, or heel.
3. 2D Photographs of both feet will be performed for a visual baseline assessment skin and soft tissue thickness.

If the clinical fat graft procedure occurs on a day different from the screening visit, the following research activities will be completed at Visit 2 if the subject continues to remain interested and eligible for study participation:

1. Collection of subject's vital signs (Temp, HR, Resp., BP), medication profile, allergies, weight, BMI calculation and adverse event collection and reporting.
2. Medical and surgical history collection review - the Investigator will confirm that the subject's medical status has not changed since last seen and the subject continues to satisfy eligibility criteria for study intervention.
3. Performance of a limited physical and foot exam by PI and /or Co-investigator MD
4. Women of childbearing potential will receive a urine pregnancy dip test with results documented to study chart.
5. Diary cards with instruction to start entry on the diary card 24 hours after the fat grafting surgery to continue through Post-operative Visit 4 (Month 1) and be placed to study chart. The subject will be instructed to document self-assessment of the following events pertaining to the surgical site: Pain, Bruising, Redness of the skin, Itching, Swelling, Bleeding, Other (any concerns/issues not listed). The subject will be instructed to identify on the diary card the location, date and day of each documented event. Unresolved events at Visit 4 will be carried over for documentation to the adverse event log.
6. 2D Photographs of both feet
7. Offload Device Distribution to remain in use at all times during ambulation and activity instruction to stay off of feet as much as possible for 3 days, then limit ambulation to 10 minutes per hour for 4 weeks and no sports, kicking, running or exercise for 4 weeks. Devices will be provided for both feet to maintain symmetry and gait stability between the two feet.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent
2. Subjects scheduled to undergo a standard of care treatment with fat grafting for foot pain due to forefoot or heel fat pad atrophy or chronic plantar fasciitis as defined by heel pain for greater than 6 months and failed non-surgical therapy
3. Willing and able to comply with follow up examinations, including ultrasounds

Exclusion Criteria:

1. Concurrent injury to the lower extremity that would effect gait
2. Open foot ulcerations, fractures, or diagnosis of osteomyelitis of the feet
3. Surgical foot intervention in the last 6 months
4. Diagnosis of pregnancy or the intent of the participant to become pregnant during participation in this study
5. Any issue that per the physician's determination would render the patient not appropriate to continue participation in the study (compliance, change in physical status, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonography | at screening
  Tissue thickness (skin, soft tissue, and plantar fascia thickness) as assessed by ultrasound
Ultrasonography | 1 month post-op
  Tissue thickness (skin, soft tissue, and plantar fascia thickness) as assessed by ultrasound
Ultrasonography | 2 months post-op
  Tissue thickness (skin, soft tissue, and plantar fascia thickness) as assessed by ultrasound
Ultrasonography | 6 months post-op
  Tissue thickness (skin, soft tissue, and plantar fascia thickness) as assessed by ultrasound
American Orthopedic Foot and Ankle Society questionnaire (AOFAS). | at screening
  This survey assesses gait (no abnormality to severe abnormality), ankle motion restriction (no restriction to severe restriction), difficulty with waling on uneven surfaces (no difficulty to severe difficulty) and alignment (good to poor). There is no overall summation of results
American Orthopedic Foot and Ankle Society questionnaire (AOFAS). | 1 month post-op
  This survey assesses gait (no abnormality to severe abnormality), ankle motion restriction (no restriction to severe restriction), difficulty with waling on uneven surfaces (no difficulty to severe difficulty) and alignment (good to poor). There is no overall summation of results
American Orthopedic Foot and Ankle Society questionnaire (AOFAS). | 2 months post-op
  This survey assesses gait (no abnormality to severe abnormality), ankle motion restriction (no restriction to severe restriction), difficulty with waling on uneven surfaces (no difficulty to severe difficulty) and alignment (good to poor). There is no overall summation of results
American Orthopedic Foot and Ankle Society questionnaire (AOFAS). | 6 months post-op
  This survey assesses gait (no abnormality to severe abnormality), ankle motion restriction (no restriction to severe restriction), difficulty with waling on uneven surfaces (no difficulty to severe difficulty) and alignment (good to poor). There is no overall summation of results
Pittsburgh Foot Survey | at screening
  Pain and function questionnaire measure. Scale for pain ranges from "Very severe" to "Had no pain". Scale for pain interference ranges from " Very much" to "not at all". Scale of functionality ranges from "unable to do" to "without any difficulty" in regards to a range of specified activities. There is no overall summation of results
Pittsburgh Foot Survey | 1 month post-op
  Pain and function questionnaire measure. Scale for pain ranges from "Very severe" to "Had no pain". Scale for pain interference ranges from " Very much" to "not at all". Scale of functionality ranges from "unable to do" to "without any difficulty" in regards to a range of specified activities. There is no overall summation of results
Pittsburgh Foot Survey | 2 months post-op
  Pain and function questionnaire measure. Scale for pain ranges from "Very severe" to "Had no pain". Scale for pain interference ranges from " Very much" to "not at all". Scale of functionality ranges from "unable to do" to "without any difficulty" in regards to a range of specified activities. There is no overall summation of results
Pittsburgh Foot Survey | 6 months post-op
  Pain and function questionnaire measure. Scale for pain ranges from "Very severe" to "Had no pain". Scale for pain interference ranges from " Very much" to "not at all". Scale of functionality ranges from "unable to do" to "without any difficulty" in regards to a range of specified activities. There is no overall summation of results
Manchester Foot and Ankle Disability Index | at screening
  Pain and function questionnaire assessment. Three responses to a variety of pain and specified activities raging from "On most/every day(s)" which is scored as 2 to "none of the time" which is scored as 0. Summation is made on Functional (0-20 with 20 being the lowest functioning), Personal appearance (0-4 with 4 being the worst), pain (0-10 with 10 being the worst), work/leisure (0-100 with 100 being the worst impact on work/leisure).
Manchester Foot and Ankle Disability Index | 1 month post-op
  Pain and function questionnaire assessment. Three responses to a variety of pain and specified activities raging from "On most/every day(s)" which is scored as 2 to "none of the time" which is scored as 0. Summation is made on Functional (0-20 with 20 being the lowest functioning), Personal appearance (0-4 with 4 being the worst), pain (0-10 with 10 being the worst), work/leisure (0-100 with 100 being the worst impact on work/leisure).
Manchester Foot and Ankle Disability Index | 2 months post-op
  Pain and function questionnaire assessment. Three responses to a variety of pain and specified activities raging from "On most/every day(s)" which is scored as 2 to "none of the time" which is scored as 0. Summation is made on Functional (0-20 with 20 being the lowest functioning), Personal appearance (0-4 with 4 being the worst), pain (0-10 with 10 being the worst), work/leisure (0-100 with 100 being the worst impact on work/leisure).
Manchester Foot and Ankle Disability Index | 6 months post-op
  Pain and function questionnaire assessment. Three responses to a variety of pain and specified activities raging from "On most/every day(s)" which is scored as 2 to "none of the time" which is scored as 0. Summation is made on Functional (0-20 with 20 being the lowest functioning), Personal appearance (0-4 with 4 being the worst), pain (0-10 with 10 being the worst), work/leisure (0-100 with 100 being the worst impact on work/leisure).
Mayo Clinical Scoring System questionnaire (MAYO) | at screening
  Pain and function questionnaire. Pain scale from 0 (worst) to 50 (no pain). Activity limitations, orthotic requirements, antalgic gait, neuropathy and plantar heel tenderness are all graded 10 (best) to 10 (worst). Overall summation is excellent (90-100), good (80-89), fair (70-79), poor (<70)
Mayo Clinical Scoring System questionnaire (MAYO) | 1 month post-op
  Pain and function questionnaire. Pain scale from 0 (worst) to 50 (no pain). Activity limitations, orthotic requirements, antalgic gait, neuropathy and plantar heel tenderness are all graded 10 (best) to 10 (worst). Overall summation is excellent (90-100), good (80-89), fair (70-79), poor (<70)
Mayo Clinical Scoring System questionnaire (MAYO) | 2 months post-op
  Pain and function questionnaire. Pain scale from 0 (worst) to 50 (no pain). Activity limitations, orthotic requirements, antalgic gait, neuropathy and plantar heel tenderness are all graded 10 (best) to 10 (worst). Overall summation is excellent (90-100), good (80-89), fair (70-79), poor (<70)
Mayo Clinical Scoring System questionnaire (MAYO) | 6 months post-op
  Pain and function questionnaire. Pain scale from 0 (worst) to 50 (no pain). Activity limitations, orthotic requirements, antalgic gait, neuropathy and plantar heel tenderness are all graded 10 (best) to 10 (worst). Overall summation is excellent (90-100), good (80-89), fair (70-79), poor (<70)
Foot and Ankle Ability Measure (FAAM) questionnaire | at screening
  Mobility and functionality questionnaire. Scale ranges from "Unable to do" to "no difficulty at all" in response to questions on mobility. There is no overall summation of results.
Foot and Ankle Ability Measure (FAAM) questionnaire | 1 month post-op
  Mobility and functionality questionnaire. Scale ranges from "Unable to do" to "no difficulty at all" in response to questions on mobility. There is no overall summation of results.
Foot and Ankle Ability Measure (FAAM) questionnaire | 2 months post-op
  Mobility and functionality questionnaire. Scale ranges from "Unable to do" to "no difficulty at all" in response to questions on mobility. There is no overall summation of results.
Foot and Ankle Ability Measure (FAAM) questionnaire | 6 months post-op
  Mobility and functionality questionnaire. Scale ranges from "Unable to do" to "no difficulty at all" in response to questions on mobility. There is no overall summation of results.

SECONDARY OUTCOMES:
Offload Device Survey | at screening
  Device satisfaction measure questionnaire. Questions are answered yes/no in all cases except comfort (0-10 with 10 being the most comfortable), ease of use (0-10 with 10 being most easy to use) and how many hours per night a patient needed to wear a night splint (0-8).
Offload Device Survey | 2 weeks post-op
  Device satisfaction measure questionnaire. Questions are answered yes/no in all cases except comfort (0-10 with 10 being the most comfortable), ease of use (0-10 with 10 being most easy to use) and how many hours per night a patient needed to wear a night splint (0-8).
Offload Device Survey | 1 month post-op
  Device satisfaction measure questionnaire. Questions are answered yes/no in all cases except comfort (0-10 with 10 being the most comfortable), ease of use (0-10 with 10 being most easy to use) and how many hours per night a patient needed to wear a night splint (0-8).
Offload Device Survey | 2 months post-op
  Device satisfaction measure questionnaire. Questions are answered yes/no in all cases except comfort (0-10 with 10 being the most comfortable), ease of use (0-10 with 10 being most easy to use) and how many hours per night a patient needed to wear a night splint (0-8).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Gusenoff, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee Women's Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No